CLINICAL TRIAL: NCT01243281
Title: A Randomized Design Study to Compare the Efficacy of Pegylated Interferon Alpha-2b Monotherapy Versus Combination With Entecavir in HBeAg-negative Chronic Hepatitis B: Role of Host and Viral Factors Associated With Treatment Response
Brief Title: Pegylated Interferon Alpha-2b Monotherapy Versus Combination With Entecavir in HBeAg-negative Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Dr. Pisit Tangkijvanich, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biochem2010/01
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis B
Keywords: hepatitis B; HBeAg; pegylated interferon; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir; peginterferon alfa-2b

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug combination (Active Comparator)
  Interventions: Drug: PEG-IFN and entecavir

INTERVENTIONS:
Drug: PEG-IFN and entecavir — The patients will be randomized in approximately 1:1 ratio into one of 2 treatment regimens; to receive PEG-IFN alpha-2b (1.5 microgram/kg/week) plus entecavir (0.5 mg/day) or PEG-IFN alpha-2b (1.5 microgram/kg/week) alone for 48 weeks by using pre-generated randomization schedule.
  Other Names: pegintron; baraclude

SUMMARY:
The outcome of treatment of chronic hepatitis B is determined by viral and host interaction, thus the combination therapy of immunomodulator (PEG-IFN) and potent antiviral drug (entecavir) should improve the response rate. In addition, the simultaneous assessment of viral and host genetic factors associated with SVR may help to identify predictors of treatment outcomes, which will in turn significant reduce the cost/effect of therapy

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age
* Patients with HBeAg-negative chronic hepatitis B
* Positive for HBsAg for at least 6 months, negative for anti-HBs and HBeAg
* Serum HBV DNA levels ≥ 2,000 IU/mL at screening
* Increased alanine aminotransferase (ALT) levels [greater than the upper limit of normal (ULN) and less than 10xULN}
* No signs or symptoms of advanced liver disease
* Patient has had a liver biopsy within 1 year of screening

Exclusion Criteria:

* Patient had previous treatment with IFN, peg-IFN, and/or entecavir
* Patient has evidence or history of chronic hepatitis not caused by HBV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis
* Patient has co-infection with hepatitis C virus and/or human immunodeficiency virus
* Patients with liver cancer
* Female patient is pregnant, lactating, expecting to conceive or donate eggs, or is of childbearing potential throughout treatment.
* Patient has any other condition that is contraindicated for treatment with PEG-IFN or entecavir
* Patient has any condition or pre-study laboratory abnormality, or history of any illness, which in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether a combination of PEG-IFN and entecavir improves the rate of sustained response and HBsAg clearance in patients with HBeAg-negative chronic hepatitis B | 24 weeks post treatment

SECONDARY OUTCOMES:
To determine host factors and viral factors associated with response to PEG-IFN alone or PEG-IFN plus entecavir treatment | 24 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pisit Tangkijvanich, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand